CLINICAL TRIAL: NCT02740543
Title: Biomarkers of Irritant-Induced and Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-01191
Record Dates: First submitted 2016-04-08; First posted 2016-04-15 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Asthma
Keywords: World Trade Center; WTC; Induced Sputum; Exhaled Breath Condensate
MeSH Terms: conditions — Asthma | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergic Asthma (AA) (Active Comparator)
  Interventions: Drug: Fluticasone propionate HFA 220
- Control (No Intervention)

INTERVENTIONS:
Drug: Fluticasone propionate HFA 220 — Subjects will take two (2) puffs of Fluticasone propionate HFA 220 twice a day.
  Other Names: Corticosteroid
  Arms: Allergic Asthma (AA)

SUMMARY:
Asthma is a heterogeneous disease, and although much is understood about mechanisms of inflammation in allergic asthma, less is known about mechanisms of irritant-induced asthma (IA). Understanding the underlying similarities and differences in mechanisms of these two types of asthma will help focus current treatments and lead to development of new therapies. There is a longstanding NYU/Bellevue Asthma registry (NYUBAR), with a large population (N = 900) of asthma cases and controls, a program that has been housed at the CTSI (formerly GCRC). The destruction of the World Trade Center (WTC) resulted in massive dust, gas and fume exposures to local residents, workers and cleanup workers and individuals involved in rescue and recovery and adverse respiratory health effects of this disaster are reported more than 7 years after 9/11. Many responders, as well as those exposed as residents or local workers, have developed IA, asthma that arises after a lag from an environmental exposure . The WTC Environmental Health Center (WTC EHC) is one of the three New York City (NYC) WTC Centers of Excellence and the only one that focuses on treatment and monitoring of local workers and residents. As such, it has a large population of individuals with irritant-induced asthma. It has been proposed to use participants from the NYUBAR and the WTC EHC to expand the knowledge of irritant and allergic asthma. Non-invasive studies allow for the assessment of airway inflammation, a non-specific response to environmental exposure and injury. Recent technologies also allow for assessment of microRNA (miRNA), small RNAs that regulate gene expression at the post-transcriptional level and thus serve as a pathway to regulation of inflammation. The hypothesis will be tested in that airway inflammation in irritant and allergic asthma may be similar, but result from divergent miRNA regulatory pathways expressed in sputum cells. These studies will provide preliminary data for future studies that will help identify biological pathways to categorize these asthma phenotypes and target future treatment interventions.

DETAILED DESCRIPTION:
This study will have two asthma phenotypes and one control population. Patients will be recruited from the WTC EHC = 30 with WTC dust cloud exposure, patients will be recruited from the NYUBAR (n=30) and have asthma as defined by NIH guidelines, and control patients will be recruited from the NYUBAR (n=30) and will have no respiratory sx, no asthma diagnosis, or no WTC dust exposure.

The study will entail two to three visits. On visit 1 (V1) all individuals will sign informed consent to participate in the study under an NYU IRB approved protocol. A questionnaire will be completed with standardized questions that include information on WTC exposures, demographics, presence and severity of respiratory symptoms, tobacco history and past medical history. Individuals will undergo spirometry with inhaled bronchodilator. Individuals will undergo methacholine challenge test (visit 1a) if they have normal spirometry or no bronchial hyperresponsiveness. On visit 2, individuals will return to undergo ENO, EBC and spirometry with pre and post bronchodilator maneuvers and induced sputum. Blood will be obtained for CBC with differential cell count, and assessment of total IgE and allergen-specific IgE. Blood will also be stored for future analysis of inflammatory markers. Based on experience, there have been individuals unable to produce enough sputum and thus yield too small a number of cells. These individuals are excluded from data analysis. In addition, there will also be subjects who are able to produce sputum and return for repeat sputum testing.

ELIGIBILITY:
Inclusion Criteria:

For the WTC population with Irritant-Induced Asthma (IA):

* > 18 years of age*
* Current nonsmoker*
* < 5 pack year (p-y) history of tobacco use*
* Spirometry in the past 6 months or on day of evaluation with a bronchodilator* response of ≥ 12% and 200 ml improvement in FEV*
* Positive methacholine challenge test (decrease in FEV1*

  ≥ 20% (PC20) after inhalation of < 16 mg/ml of methacholine)
* Inhaled corticosteroid use in previous 1 month or more will be allowed*
* Patients will be recruited from the WTC EHC and will have WTC dust cloud exposure
* New symptoms after 9/11
* Symptoms of wheeze and shortness of breath (> 2x / week) in the 4 weeks before inclusion (persistent symptoms).

Inclusion for Allergic Asthma Population (AA):

* All of the above items with an asterisk (*)
* Patients will be recruited from the NYUBAR or advertisement and will have asthma as defined by NIH guidelines, persistent symptoms, absence of WTC dust exposure.
* Participants who will have completed the Phase I of the study and were able to produce adequate sputum samples.

Inclusion of Control Population:

* Patients will be recruited from the NYUBAR and will have no respiratory symptoms, no asthma diagnosis, no WTC dust exposure, no current tobacco use, ≤ 5 p-y history of tobacco use, and normal spirometry with no bronchodilator response and negative methacholine challenge in past 6 months.

Inclusion Criteria for Phase II:

* Successfully completed Phase I
* Has asthma according to Phase I diagnostic criteria
* Signed consent to be re-contacted

Exclusion Criteria:

* Current Smoker
* Pulmonary diseases such as Chronic Pulmonary Disease (COPD) or Interstitial Lung Disease
* Cardiac Disease
* Inability to perform lung function or other maneuvers
* Upper respiratory tract infection within the last 4 weeks
* FEV1 <60% predicted normal pre-bronchodilator
* Oral corticosteroid treatment within the last 4 weeks.
* No vulnerable subjects will be part of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Kazeros, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No fluticasone propionate HFA was given to participants.
Period: Overall Study
Arm/Group | Allergic Asthma (AA) | Control
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergic Asthma (AA) | Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (7) | 33 (8) | 30 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in TSLP Gene Expression
Description: The primary outcome is the change in TSLP gene expression in epithelial cells after 2 weeks of treatment of inhaled corticosteroid compared to no treatment.
Time Frame: Baseline and Two (2) weeks
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Allergic Asthma (AA) | Control
Number analyzed (Participants) | 9 | 9
Fold Change | 0.000197 (0.000134) | 0.000035 (0.000023)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Control: Fluticasone propionate HFA was not given to participant
Arm/Group | Allergic Asthma (AA) | Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02740543/Prot_SAP_000.pdf